CLINICAL TRIAL: NCT03408262
Title: A Phase I Single-Blind Randomised Trial Investigating Immunisation Strategies Using Ad4-EnvCN54, MVA-CN54 and CN54gp140/MPLA Combinations in Order to Maximise Antibody Responses to Human Immunodeficiency Virus
Brief Title: Clinical Trial of HIV Vaccine Combinations in Healthy Men and Women
Acronym: Ad4HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ad4HIV
Record Dates: First submitted 2018-01-05; First posted 2018-01-23 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Group A (Active Comparator): Month 0: oral placebo Month 3: oral placebo + I.M. CN54gp140/MPLA + I.M. placebo Month 6: oral placebo + I.M. CN54gp140/MPLA + I.M. placebo
  Interventions: Biological: CN54gp140/MPLA
- Group B (Experimental): Month 0: Ad4-EnvCN54 Month 3: oral placebo + I.M. CN54gp140/MPLA + I.M. placebo Month 6: oral placebo + I.M. CN54gp140/MPLA + I.M. placebo
  Interventions: Biological: Ad4-EnvCN54; Biological: CN54gp140/MPLA
- Group C (Experimental): Month 0: Ad4-EnvCN54 Month 3: Ad4-EnvCN54 + I.M. CN54gp140/MPLA + I.M. placebo Month 6: oral placebo + I.M. CN54gp140/MPLA + I.M. placebo
  Interventions: Biological: Ad4-EnvCN54; Biological: CN54gp140/MPLA
- Group D (Experimental): Month 0: Ad4-EnvCN54 Month 3: Ad4-EnvCN54 + I.M. CN54gp140/MPLA + I.M. placebo Month 6: Ad4-EnvCN54 + I.M. CN54gp140/MPLA + I.M. placebo
  Interventions: Biological: Ad4-EnvCN54; Biological: CN54gp140/MPLA
- Group E (Active Comparator): Month 0: oral placebo Month 3: oral placebo + I.M. CN54gp140/MPLA + I.M. MVA-CN54 Month 6: oral placebo + I.M. CN54gp140/MPLA + I.M. MVA-CN54
  Interventions: Biological: MVA-CN54; Biological: CN54gp140/MPLA
- Group F (Experimental): Month 0: Ad4-EnvCN54 Month 3: oral placebo + I.M. CN54gp140/MPLA + I.M. MVA-CN54 Month 6: oral placebo + I.M. CN54gp140/MPLA + I.M. MVA-CN54
  Interventions: Biological: Ad4-EnvCN54; Biological: MVA-CN54; Biological: CN54gp140/MPLA
- Group G (Experimental): Month 0: Ad4-EnvCN54 Month 3: Ad4-EnvCN54 + I.M. CN54gp140/MPLA + I.M. MVA-CN54 Month 6: oral placebo + I.M. CN54gp140/MPLA + I.M. MVA-CN54
  Interventions: Biological: Ad4-EnvCN54; Biological: MVA-CN54; Biological: CN54gp140/MPLA
- Group H (Experimental): Month 0: Ad4-EnvCN54 Month 3: Ad4-EnvCN54 + I.M. CN54gp140/MPLA + I.M. MVA-CN54 Month 6: Ad4-EnvCN54 + I.M. CN54gp140/MPLA + I.M. MVA-CN54
  Interventions: Biological: Ad4-EnvCN54; Biological: MVA-CN54; Biological: CN54gp140/MPLA

INTERVENTIONS:
Biological: Ad4-EnvCN54 — Live, replication-competent adenovirus 4 vector, engineered to express the envelope glycoprotein of HIV-1 isolate 97CN54
  Arms: Group B; Group C; Group D; Group F; Group G; Group H
Biological: MVA-CN54 — Live, non-replicating modified vaccinia Ankara vector, engineered to express the envelope glycoprotein of HIV-1 isolate 97CN54
  Arms: Group E; Group F; Group G; Group H
Biological: CN54gp140/MPLA — Recombinant glycoprotein of HIV-1 isolate 97CN54, with liposomal monophosphoryl lipid A adjuvant
  Other Names: CN54-M

SUMMARY:
A Phase I Single-Blind randomised trial investigating immunisation strategies using Ad4-EnvCN54, MVA-CN54 and CN54gp140/MPLA combinations in order to maximise antibody responses to Human Immunodeficiency Virus

DETAILED DESCRIPTION:
This is a randomised two-part Phase I study which will explore the impact of different boosting options (MVA-CN54 and recombinant CN54gp140 protein) for oral Adenovirus serotype 4 vector prime expressing HIV-1 CN54 envelope (Ad4-EnvCN54) designed to optimize systemic and mucosal antibody responses.

Part 1 is exploratory and designed to select conditions capable of promoting enhanced systemic and mucosal B cell responses in a limited number of participants.

Part 2 is dependent upon Part 1 and is designed to study groups selected on performance in part 1 in an expanded number of subjects. Data from both stages will be combined for safety and immunological analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 18 and 50 years on the day of screening
2. BMI between 18-30
3. Seronegative for Adenovirus 4 serum neutralising antibodies
4. Available for follow-up for the duration of the study
5. Willing and able to give written informed consent
6. At low risk of HIV infection and willing to remain so for the duration of the study defined as:

   * no history of injecting drug use in the previous ten years
   * no gonorrhoea or syphilis in the last six months
   * no high risk partner (e.g. injecting drug use, HIV positive partner) either currently or within the past six months
   * no unprotected anal or vaginal intercourse in the last six months, outside a relationship with a regular partner known to be HIV negative
7. Willing to undergo HIV testing
8. Willing to undergo a STI screen for chlamydia, gonorrhoea and syphilis
9. Must agree to require male sexual partner to use condoms, from at least 14 days before the first vaccination until at least 4 months after the last
10. If heterosexually active female capable of becoming pregnant, must (in addition to requiring male partner to use condoms) agree to use hormonal contraception, or to complete abstinence, from at least 30 days before the first vaccination until at least 4 months after the last. [Note: Acceptable hormonal contraception is combined (estrogen and progestogen containing) or progestogen-only hormonal contraception associated with inhibition of ovulation. Complete abstinence can be used, when in line with the preferred and usual lifestyle of the subject. Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, lactational amenorrhoea method, and IUD/IUS are not acceptable methods of contraception.]
11. If sexually active male, must agree to use condoms from the day of first vaccination until at least 4 months after the last. [Note: Additional use of an effective method of contraception is recommended for any non-pregnant female partner over the same period.]
12. Agree to abstain from donating blood, eggs or sperm from the day of first vaccination until at least 3 months after the end of their participation in the trial
13. Registered with a GP for at least the past month
14. Entered and clearance obtained from The Overvolunteering Prevention System (TOPS) database

Exclusion Criteria:

1. Are pregnant or breast feeding, or living with anyone under the age of 5 years old or over 75 years old
2. Have close contact with an immunocompromised individual thought to be at clinical risk from Adenovirus infection
3. Clinically relevant abnormality on history or examination including:

   1. Liver disease with inadequate hepatic function
   2. Any skin condition which may interfere with the trial assessment of the injection sites
   3. Haematological, metabolic, gastrointestinal or cardio-pulmonary disorders
   4. Uncontrolled infection; autoimmune disease, immunodeficiency
4. Known hypersensitivity to any component of the vaccine formulations used in this trial, or have severe or multiple allergies to drugs or pharmaceutical agents
5. History of severe local or general reaction to vaccination defined as

   * Local: extensive, indurated redness and swelling involving most of the antero-lateral thigh or the arm, not resolving within 72 hours
   * General: fever ≥39.5oC within 48 hours; anaphylaxis; bronchospasm; laryngeal oedema; collapse; convulsions or encephalopathy within 72 hours
6. Receipt of live attenuated vaccine within 60 days or other vaccine within 30 days of enrolment
7. Receipt of an experimental vaccines containing HIV antigens, Ad4 and MVA-C products at any time in the past
8. Receipt of blood products or immunoglobin within 4 months of screening, or drugs that suppress the immune system, such as steroids (including inhaled steroids, excluding topical steroids unless applied to the upper arm), in the preceding 3 months
9. Participating in another trial of a medicinal product, completed less than 30 days prior to enrolment
10. HIV 1 or 2 positive or indeterminate on screening
11. Positive for antibodies to hepatitis B surface antigen, hepatitis C antibody or serology indicating active syphilis requiring treatment
12. Clinically significant positive reaction in antinuclear antibody screen or clinically significant immunoglobulin (IgA, IgG or IgM) values
13. Grade 1 or above clinically significant routine laboratory parameters
14. Unable to read and/or speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent
15. Women with a history of toxic shock syndrome
16. Women using an intrauterine device for contraception (as incompatible with softcup sampling)
17. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
18. Unlikely to comply with protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Lewis, MD, Principal Investigator — Imperial College London
Locations (1):
- NIHR Imperial Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Group G | Group H
Started | 15 | 6 | 6 | 13 | 6 | 6 | 9 | 7
Completed | 11 | 6 | 6 | 12 | 6 | 6 | 6 | 6
Not Completed | 4 | 0 | 0 | 1 | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Healthy male or female adults, 18 to 50 years of age, at low risk for HIV infection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Group G | Group H | Total
Number analyzed (Participants) | 15 | 6 | 6 | 13 | 6 | 6 | 9 | 7 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 6 | 6 | 13 | 6 | 6 | 9 | 7 | 68
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 3 | 6 | 2 | 2 | 4 | 3 | 29
  Male | 8 | 4 | 3 | 7 | 4 | 4 | 5 | 4 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 7 | 3 | 3 | 3 | 2 | 5 | 4 | 1 | 28
  White Irish | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any other white background | 5 | 0 | 0 | 3 | 4 | 0 | 2 | 3 | 17
  Indian | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 4
  Pakistani | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Bangladeshi | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any other Asian background | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 6
  Mixed White and Black Caribbean | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Mixed White and Black African | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Mixed White and Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any other Mixed background | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Black Caribbean | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3
  Black African | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 4
  Any other Black background | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15 | 6 | 6 | 13 | 6 | 6 | 9 | 7 | 68
Number of participants with CN54-gp140 IgG antibodies at time of vaccination [Count of Participants; unit: Participants] — CN54-gp140 serum IgG antibodies were measured at baseline, before the participants received any vaccinations
  Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Mucosal Binding IgG Antibodies to HIV CN54gp140 Antigen
Description: Number of participants with mucosal (semen, nasal, vaginal or rectal) binding IgG antibodies to HIV CN54gp140 antigen, as determined by ELISA
Time Frame: At two weeks after the final immunisation
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Group G | Group H
Number analyzed (Participants) | 11 | 6 | 6 | 12 | 6 | 6 | 6 | 6
Participants | 0 | 3 | 1 | 6 | 0 | 1 | 2 | 1

2. Primary Outcome: Number of Participants With Severe or Greater (Grades 3-4) Adverse Reactions During the Study
Description: Number of Participants With Severe or Greater (Grades 3-4) Adverse Reactions up to twenty-four weeks after the final immunisation
Time Frame: Up to twenty-four weeks after the final immunisation
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Group G | Group H
Number analyzed (Participants) | 15 | 6 | 6 | 13 | 6 | 6 | 9 | 7
Participants | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3

3. Primary Outcome: Median Concentration of CN54-gp140 Specific IgG Binding Antibodies
Description: Median concentration of CN54-gp140 specific IgG binding antibodies, as measured by ELISA. Concentration is in ng/mL
Time Frame: At two weeks after the final immunisation
Population: Serum from participants at two weeks after the final immunisation
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Group G | Group H
Number analyzed (Participants) | 7 | 6 | 6 | 9 | 6 | 6 | 6 | 6
ng/mL | 464 [23 to 1521] | 14141 [3971 to 18348] | 8992 [3798 to 79435] | 11367 [398 to 26149] | 6280 [1102 to 15044] | 9639 [3250 to 14282] | 20512 [10583 to 36552] | 9041 [4735 to 21023]

4. Secondary Outcome: Number of Participants With Detectable Serum Binding Antibodies to HIV CN54gp140 Antigen
Description: Number of participants with detectable serum binding antibodies to HIV CN54gp140 antigen, as measured by IgG binding ELISA
Time Frame: At two weeks post-final immunisation
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Group G | Group H
Number analyzed (Participants) | 11 | 6 | 6 | 12 | 6 | 6 | 6 | 6
Participants | 7 | 6 | 5 | 11 | 6 | 6 | 6 | 6

ADVERSE EVENTS:
Time Frame: 12 months
Description: All adverse events were recorded. Grades were defined as 1 (mild), 2 (moderate), 3 (severe) or 4 (life threatening).
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Group G | Group H
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/6 | 1/6 | 0/12 | 0/6 | 1/6 | 0/6 | 3/6
Other Adverse Events (participants affected / at risk) | 6/12 | 3/6 | 2/6 | 9/12 | 3/6 | 3/6 | 3/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=12) | Group B (N=6) | Group C (N=6) | Group D (N=12) | Group E (N=6) | Group F (N=6) | Group G (N=6) | Group H (N=6)
Depressive Disorder Triggering Overdose (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTI on Kidney stones (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis secondary to Mallory Weiss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis on hand (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=12) | Group B (N=6) | Group C (N=6) | Group D (N=12) | Group E (N=6) | Group F (N=6) | Group G (N=6) | Group H (N=6)
Myalgia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenderness left arm (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (3) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Right wrist synovialcyst surgical removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea/nasopharyngitis/rhinitis/cold/upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 2 (2) | 2 (4) | 4 (4) | 1 (2) | 1 (1) | 3 (4) | 1 (1)
Road traffic accident (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sports injury (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lateral femoral nerve compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting, vision blurred, headache and fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hangover/Alcoholic Withdrawal Symptoms (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feverish (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dygeusia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biceps tendon tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
shoulder/clavicle region tenderness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Threadworm infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT03408262/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT03408262/SAP_001.pdf